CLINICAL TRIAL: NCT05612997
Title: Relative Validation of a Remote Novel Food Frequency Questionnaire Compared to 24hr Recalls in the ZOE AFFIRM Study
Brief Title: ZOE-AFFIRM: Relative Validation of a Novel Food Frequency Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: Zoe Global Limited (Other)
Responsible Party: Sponsor
Other Study IDs: ZOE-AFFIRM
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relative Validation Arm
  Interventions: Other: Dietary Assessment

INTERVENTIONS:
Other: Dietary Assessment — Food Frequency Questionnaire and 24h Recalls.

SUMMARY:
Dietary assessment is critical for dietary research. Food Frequency Questionnaires (FFQ) measure habitual dietary intake and are low user and researcher burden. The ZOE AFFIRM study aims to assess the relative validity of a novel FFQ compared to a widely accepted 24h dietary recall tool in a remote setting.

DETAILED DESCRIPTION:
Research Question:

What is the relative validity of a novel FFQ (Food Frequency Questionnaire) compared to a widely accepted 24h dietary recall tool in a remote setting?

Research Aim:

This study aims to relatively validate the ZFFQ (ZOE Food Frequency Questionnaire; ZOE Ltd) by assessing its agreement with a widely accepted 24h diet recall tool, Intake24 (Newcastle University) in a remote population.

Design:

This study will be conducted in a single-arm design with the intake period under assessment comprising one month.

1. Participants will complete two periods of 3 consecutive days each (one weekend-day and two weekdays, i.e. Sunday-Tuesday or Thursday-Saturday), in which they will complete 6 total rounds of Intake24 (one completion per previous 24 hours). The two periods must be at least 14 days apart; participants will be given multiple options of dates to choose from in November/December that satisfy these requirements.
2. Once the two recall periods are completed, the participant will be asked to fill out the ZFFQ recalling food frequency (without portion sizes) over the preceding month (which encompasses the two recall periods).

Population: In brief, participants are generally healthy UK-based adults who provided consent to participation in this remote study. Please see the eligibility section for full criteria. Participants provided consent before undertaking any study procedures.

Data analysis: Agreement analysis will be used to compare both dietary assessment methods and evaluate the relative validity of the ZOE FFQ.

Data collection:

* Baseline demographic data (age, sex, BMI, ethnicity, smoking, socio-economic status)
* Dietary data (FFQ and 24hr dietary recall)

ELIGIBILITY:
Inclusion Criteria:

* Can provide written informed consent
* Are willing and able to comply with all study protocols
* Are willing to complete their dietary recall periods on specified dates
* Have BMI 18 and above
* Are any sex
* Are aged 18 years old and above
* Live in England, Scotland, Wales or Northern Ireland

Exclusion Criteria:

- Do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: United Kingdom-based adult population who have subscribed to the ZOE Product waitlist.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-11-08 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Food Frequency Questionnaire | 30 days
24h Recalls | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Berry, PhD, Principal Investigator — King's College London and Consultant at ZOE Ltd
Locations (1):
- ZOE Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No